CLINICAL TRIAL: NCT05342441
Title: Optimizing GRAft SElection for ACL Reconstruction (GRASE-ACL Trial) - a Three-armed Randomized Controlled Trial
Brief Title: Optimizing Graft Selection for ACL Reconstruction
Acronym: GRASE-ACL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University College Copenhagen (Other); National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Kristoffer Barfod, Consultant, MD, PhD, Associate Professor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRASE ACL
Record Dates: First submitted 2022-04-04; First posted 2022-04-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
Keywords: ACL reconstruction; Graft choice; Quadriceps graft; Semitendinosus/gracilis graft; Muscle morphology; Neuromuscular control; BPTB graft; Patient reported function
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Prospective, assesor blinded randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Before each patient visit, tape will be placed on possible scars to hide donor graft site. Given the nature of the intervention, blinding of patients and surgeons is not feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QT-graft (Experimental): Quadriceps tendon autograft (n=50)
  Interventions: Procedure: QT graft
- St/Gr-graft (Experimental): Semitendinosus/gracilis autograft (n=50)
  Interventions: Procedure: ST/Gr graft
- BPTB-graft (Experimental): Patella tendon autograft (n=50)
  Interventions: Procedure: BPTB graft

INTERVENTIONS:
Procedure: QT graft — Surgical reconstruction of primary ACL rupture with autograft harvested from the quadriceps tendon without bone block.
  The QT graft is harvested through a 4-5 cm incision at the upper pole of the patella. A graft sized 10-12 mm in with and app. 6 mm in depth is harvested from the middle part of the tendon.
  The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus.
  The ST/Gr graft is fixed proximally with the RIGIDFIX® Curve Cross Pin System (DePuy Synthes) and distally with a Milagro skrew (DePuy Synthes) or similar.
  Arms: QT-graft
Procedure: ST/Gr graft — Surgical reconstruction of primary ACL rupture with autograft harvested from the semitendinosus and gracilis muscles.
  The ST/Gr graft is harvested through a 4-5 cm incision at the pes anserinus. Both the semitendinosus and the gracilis tendon is identified and harvested. The tendons are prepared and folded to a four-stranded graft with a total diameter of 7-10 mm.
  The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus.
  The ST/Gr graft is fixed proximally with the RIGIDFIX® Curve Cross Pin System (DePuy Synthes) and distally with a Milagro skrew (DePuy Synthes) or similar.
  Arms: St/Gr-graft
Procedure: BPTB graft — Surgical reconstruction of primary ACL rupture with autograft harvested from the patella tendon with bone block (bone-patellar-tendon-bone).
  The BPTB graft is harvested through two 4-5 cm incisions, one on the tibial tuberosity and one on the patella. The middle 10 mm of the patella tendon plus 20-30 mm bone plugs at each end from corresponding tibia and patella is harvested.
  The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus. The BPTB graft is fixed both proximally and distally with a Milagro skrew (DePuy Synthes) or similar.
  Arms: BPTB-graft

SUMMARY:
Purpose:

To investigate the differences between the three most common methods for reconstruction of the anterior cruciate ligament (ACL), to support the development of the best method for the individual patient.

Main research area: ¨ Sports Orthopedic Surgical research.

State of the art:

Every year in Denmark 2500 patients receive surgical reconstruction surgery to replace a ruptured ACL. Many patients experience a decline in knee function and 4-12% suffer a new ACL rupture within 5 years. According to data from the Danish ACL register, three methods of reconstruction are most prevalent, but with large variation between hospitals. This indicates lack of consensus on optimal surgical procedure.

Design:

Assessor-blinded randomized controlled study. 150 patients aged 18-40 with ruptured ACL are allocated to reconstruction with tendon(s) harvested from either the semitendinosus and gracilis, or the patella tendon, or the quadriceps tendon. Patient follow-up will be conducted preoperatively and 1, 6, 12, 24 months postoperatively.

Primary technologies and outcomes:

* Patient-reported knee-joint function, quality of life and donor-site morbidity is obtained with standardized questionnaires. Primary outcome is subjective knee function with the International Knee Documentation Committee evaluation form (IKDC)
* Instrumented analysis of knee-joint coordination and neuromuscular control including 3-D motion capture and electromyography (EMG) during single leg jumps, landings and change-of-direction. Measurement of maximal explosive muscle power in knee extension and flexion. Primary outcome is relative difference between injured and healthy leg in rate of force development (RFD-LSI).
* Standard clinical knee examination of range of motion and instrumented examination of knee-joint stability.
* Magnetic Resonance Imaging (MRI) of the thigh muscles for examination of muscle morphology.

The trial is designed for publication in three primary publications

1. - Patient reported effect of graft choice in ACL reconstruction
2. - Biomechanical effect of graft choice in ACL reconstruction
3. - Clinical effect of graft choice in ACL reconstruction

Additional secondary publications are in the pipeline. Reference to primary protocol and results will always be emphasized in secondary publication to ensure methodological transparency.

DETAILED DESCRIPTION:
Purpose:

The aim of this randomized controlled trial is to investigate the effect of graft choice in anterior cruciate ligament (ACL) reconstruction surgery, primarily from a patient-centered as well as a novel biomechanical perspective; and secondly from a clinical and muscle morphological perspective.

The study compares the three most common methods for ACL reconstruction: autograft harvested from the m. quadriceps tendon (QT), the hamstring tendons (ST/Gr), and the patella tendon (BPTB).

By applying this 360° scientific approach, it is the hope to improve the possibilities for a much-needed evidence-based and individualized treatment of ACL ruptures.

Objectives and hypotheses:

• Objective no. 1: The patient-centered perspective To investigate the effect of graft choice on patient-reported questionnaire scores, primarily on the International Knee Documentation Committee Evaluation Form (IKDC).

The investigators hypothesize that of all three grafts, the QT graft will result in non-inferior patient reported knee function.

* Objective no. 2: The biomechanical perspective To investigate the effect of graft choice on muscle strength and knee joint control. The investigators hypothesize that of all three grafts, the ST/Gr graft will show largest negative effect on explosive muscle strength.
* Objective no. 3: The clinical perspective To explore the effect of graft choice on knee stability and surgery complications.
* Objective no. 4: The muscle morphological perspective To explore the effect of graft choice on length and cross section area of the hamstring tendons.

State-of-the-art:

The most common method for ACL reconstruction in Denmark is the use of an autograft to replace the ruptured ACL. The autograft is harvested from either the m. quadriceps tendon (QT), the m. semitendinosus and m. gracilis tendons (hamstrings) (ST/Gr), or the patella tendon with bone plugs (BPTB).

The BPTB graft was initially used as standard method. It has the advantages of faster graft incorporation (bone to bone healing), reliable graft size and low risk of graft rupture and knee laxity. It is widely used around the world. In Denmark it accounts for app. 10% of all reconstructions. A number of disadvantages of the BPTB graft have been described in the literature: anterior knee pain, pain from the donor site, extension strength deficits, and decreased knee joint flexion range of motion.

Due to these potential morbidity problems of the BPTB graft, there was a shift towards the ST/Gr graft as the preferred choice. Today, the ST/Gr graft is harvested in more than 52% of all ACL reconstructions in Denmark. From a surgeon's perspective, the graft is easy to harvest, time efficient, and leaves smaller scars. The ST/Gr graft is however associated with increased laxity of the knee joint compared to the BPTB graft, and the size of the graft can be a challenge. Also, harvest of the ST/Gr graft is associated with sustained loss of strength, length, and volume of the harvested muscles. This is of concern, as biomechanical research has shown that semitendinosus is essential to stabilize the knee joint and protect the ACL during cutting movements. Finally, recent research indicates higher risk of revision surgery using the ST/Gr graft compared to the BPTB graft.

Currently, particularly in Scandinavia, surgeons are reintroducing a third graft, the QT graft. The advantages of the QT graft are large and predictable graft size and acceptable clinical outcomes. A recent study from the Sports Orthopedic Research Center - Copenhagen (SORC-C) at Hvidovre Hospital found no difference in revision rates between the ST/Gr graft and the QT graft in a cohort of more than 400 patients. The QT graft now accounts for app. 10% of all ACL reconstructions in Denmark, but the graft remains a relatively untested method.

Methods:

Study design and approvals:

This is an assessor-blinded randomized controlled trial with a three-group parallel design. Patients will be randomized to ACL reconstruction with either BPTB, ST/Gr, or QT graft with a 1:1:1 allocation. Follow-up will be performed 1, 6, 12, and 24 months after reconstruction.

The study will adhere to the CONSORT guidelines for reporting of Multi-Arm Parallel-Group Randomized Trials (http://www.consort-statement.org) and is pre-registered at http://www.clinicaltrials.gov.

The study is approved by the Scientific Ethics Committee for the Capital Region (Journal-no.: H-19001194) and by the Danish Data Protection Agency (Jr. no. VD-2018-524)

Randomization and blinding:

Patients will be randomly assigned to a treatment group using a 1:1:1 allocation ratio using a randomization schedule of permuted blocks of random sizes. The randomization will be stratified by biological sex and age. The final randomization will be made after arthroscopic assessment of the knee and evaluation according to the in- and exclusion criteria.

Outcome assessors are blinded to group allocation. Before each patient visit, tape will be placed on possible scars to hide donor graft site. Given the nature of the intervention, blinding of patients and surgeons is not feasible.

Treatment:

The procedure is initiated with knee arthroscopy. Ligament lesions, meniscus tear, and cartilage damage are inspected and treated if indicated, and ACL remnants are removed.

The BPTB graft is harvested through two 4-5 cm incisions, one on the tibial tuberosity and one on the patella. The middle 10 mm of the patella tendon plus 20-30 mm bone plugs at each end from corresponding tibia and patella is harvested.

The ST/Gr graft is harvested through a 4-5 cm incision at the pes anserinus. Both the semitendinosus and the gracilis tendon is identified and harvested. The tendons are prepared and folded to a four-stranded graft with a total diameter of 7-10 mm.

The QT graft is harvested through a 4-5 cm incision at the upper pole of the patella. A graft sized 10-12 mm in with and app. 6 mm in depth is harvested from the middle part of the tendon.

The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus. The BPTB graft is fixed both proximally and distally with a Milagro screw (DePuy Synthes) or similar . The ST/Gr and QT grafts are fixed proximally with the RIGIDFIX® Curve Cross Pin System (DePuy Synthes) and distally with a Milagro screw (DePuy Synthes) or similar.

The patients are referred to rehabilitation according to Danish rehabilitation guidelines following ACL reconstruction.

¨

Statistics:

Analysis will be performed with a linear mixed-effects model of the relationships between outcomes and treatment group (BPTB, ST/Gr, and QT graft) and time points (pre-operative, 1-month, 6-month, 12-month, and 24-month follow-up). Fixed effects are time and treatment group, and random effects are patient ID.

Sample size:

The study includes two primary outcomes, the IKDC score change between treatment groups from pre-operative to 12-months follow-up, and the LSI-RFD between treatment groups at 12-months follow-up. The two outcomes are of different hypotheses and independent.

Based on literature, the minimal clinically important difference in IKDC score is approximately 10 points, and the standard deviation on the change in IKDC score from baseline to after ACL reconstruction is approximately 13 points. Based on these assumptions, 37 patients are needed per group (α = 0.05, β = 0.80).

A local unpublished pilot study of 10 healthy individuals showed a minimal detectable difference in LSI-RFD of 12% and a standard deviation in the group of 17%. Based on these assumptions, 40 patients are needed per group (α = 0.05, β = 0.80).

A total inclusion number of 150 is decided to account for a patient dropout of app. 10%.

ELIGIBILITY:
List of Inclusion criteria

* clinically confirmed first-time ACL rupture
* Current injury sustai´ned within 2 years
* high activity level prior to ACL rupture (Tegner score ≥ 3) and personal goal of returning to physical activity.

List of preoperative exclusion criteria

* Inadequate Danish language skills to answer questionnaires.
* Prior ligament surgery in the injured knee
* Prior ligament surgery in the non-injured knee
* Instability of the non-injured knee
* Known osteoarthritis (Kelgren Lawrence score ≥ 2)
* Prior open surgery to either knee
* Prior severe fracture involving knee joint surfaces
* Prior severe injury to thigh muscles in either leg (e.g. tear or compartment)
* Prior severe injury to the patella tendon of either knee (e.g. subluxation)
* Medical condition preventing full participation (e.g. active cancer, - rheumatoid arthritis)
* Psychiatric condition preventing full participation
* Pregnancy
* Obesity (BMI > 30)

List of Perioperative exclusion criteria (Arthroscopy)

* Medial meniscus lesion > 50%
* Lateral meniscus lesion > 50%
* Treated Meniscal root lesion or radial meniscal tear that require restrictive regimen
* Cartilage lesion >2cm2, Articular cartilage injury classification (ICRS) grade 3
* Concurrent ligament injury (except medial collateral ligament (MCL) lesion grade 1-2)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee score (IKDC). | 12 months follow up.
  Patient-reported knee function based on a questionnaire, expressed on a scale form 0-100 with 100 being the best outcome.
Rate of Torque Development - Limb Symmetry Index (RFD-LSI). | 12 months follow up
  Hamstring and quadriceps rate of torque development in the injured/operated leg compared to the healthy leg, expressed in percentage with 100% being full symmetry and the best outcome.

SECONDARY OUTCOMES:
International Knee Documentation Committee score (IKDC). | Baseline, 1, 6, and 24 months follow up.
  Patient-reported knee function based on a questionnaire, expressed on a scale form 0-100 with 100 being the best outcome.
Donor site discomfort. | Baseline, 6, 12, and 24 months follow up.
  Modified donor-site morbidity score based on the Donor-site-related functional problems questionnaire
Return to sport questionnaire. | Baseline, 6, 12 and 24 months follow up.
  Patient-reported ability, level, and performance in the sport, they want to return to following ACL reconstruction. The outcome is comparison of the qualitative data obtained in the questionnaires.
Workability questionnaire | Baseline, 1, 6, 12, and 24 months follow up.
  Patient-reported ability and disadvantages when returning to work following ACL reconstruction. The outcome is comparison of the qualitative data obtained in the questionnaires.
Patient Acceptable Symptom State questionnaire (PASS) | Baseline, 12, and 24 months.
  A patient-reported questionnaire consisting of one question regarding the patient's overall satisfaction with their knee. The outcome of the questionnaire is binary ("yes" or "no"), and the study's reported outcome is a percentage of patients who meets the threshold for PASS (provides "yes")..
Rate of torque Development - Limb Symmetry Index (RFD-LSI). | Baseline, 1, 6, and 24 months follow up.
  Hamstring and quadriceps rate of torque development in the injured/operated leg compared to the healthy leg, expressed in percentage with 100% being full symmetry and the best outcome.
Knee and hip angles. | Baseline, 6, and 12 months follow up.
  Kinematic analysis of knee and hip motion during one-legged dynamic stability exercises (balance, landing, jumping). Outcome is expressed in three-dimensional joint angles (degrees)
Knee and hip moments. | Baseline, 6, and 12 months follow up.
  Kinetic analysis of knee and hip motion during one-legged dynamic stability exercises (balance, landing, jumping). Outcome is expressed in moments (M)
Neuromuscular control. | Baseline, 6, and 12 months follow up.
  Muscle activity (EMG) during one-legged dynamic stability exercises (balance, landing, jumping).
Knee laxity | Baseline, 6, and 12 months.
  Rolimeter measurement (milimeters)
Number of patients undergoing revision surgery due to graft failure. | Baseline, 12, and 24 months follow up.
  A comparison of the number of patients undergoing revision surgery due to graft failure in each group.
Number of patients experiencing re-rupture of the operated ACL. | Baseline, 12, and 24 months follow up.
  A comparison of the number of patients experiencing re-rupture to the operated ACL in each group.
Muscle cross sectional area | At 12 months follow up.
  Hamstring and quadriceps cross sectional area expressed in square centimeters based on MRI.
Hamstring muscles retraction | At 12 months follow up.
  Hamstring muscle length expressed in centimeters based on MRI.
Number of patients experiencing rupture of the contralateral ACL. | Baseline, 12, and 24 months follow up.
  A comparison of the number of patients experiencing rupture of the contralateral ACL in each group.

OTHER OUTCOMES:
Psychological consequences | 1, 6, 12, and 24 months follow up.
  The Tampa Scale of Kinesiophobia (TSK-11). Score ranges from 11-44, where 11 means no kinesiophobia and is considered the best outcome.
Clinical knee range of motion | 6 and 12 months follow up.
  Range Of Motion (ROM) of the knee expressed in degrees from full extension to full flexion. -10 to 130 degrees is consideres normal ROM.
One-leg jump performance | 6 and 12 months follow up
  Performance in one-legged return to sport jump tests. Outcome expressed in limb symmetry of distance between injured and non-injured leg
Postoperative progress | Every second week through first year following ACL reconstruction.
  Patient-reported pain and other complications based on questionnaires via SMS-track
Postoperative rehabilitation | Every second week through first year following ACL reconstruction
  Patient-reported numbers of hours of supervised and non-supervised rehabilitation via SMS-track

CONTACTS AND LOCATIONS:
Overall Officials: Per Hölmich, D.M.Sc/D.Sc, Study Director — Hvidovre UH; Mette K Zebis, MSc, PhD, Study Director — University College Copenhagen
Locations (1):
- Copenhagen University Hospital - Amger/Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Due to national legislation on anonymisation, no raw data can be available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: By request to central contact

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT05342441/Prot_SAP_ICF_000.pdf